CLINICAL TRIAL: NCT06233721
Title: Master's Degree Graduate Nurse PhD Student
Brief Title: The Effect Of Face-To-Face and Online-Education Provided To İndividuals With Atrial Fibrillation On Medication Adherence and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Harun Küçükballı, Graduate Student, Responsible Researcher, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CUharun
Record Dates: First submitted 2023-11-29; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Oral Anticoagulant Medication; Tele-education; Medication compliance; Medication satisfaction
MeSH Terms: conditions — Atrial Fibrillation; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Control group Intervention group 1 (face-to-face education group) Intervention group 2 (tele-education group)
Who Masked: Participant, Investigator
Masking Description: Individuals who agreed to participate in the study were randomly assigned to intervention and control groups by using a randomizer (http://www.randomization.com). 150 individuals who were included in the study were randomly split into three groups by a person other than the researcher, and the three groups were given a code name. In order to generate random numbers for randomization (from 1 to 50), a software was used. Thus, determined numbers for each group were obtained. Both the participants and the researchers were blinded in group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Identifying Information Form (IIF), Medication Adherence Report Scale (MARS), and Duke Anticoagulation Satisfaction Scale (DASS) were applied to the control group two times, once in the first interview and once in the interview held a month later. The control group was not provided with education. In line with ethical principles, education and education booklet was provided to this group after the scales were applied in the last interview held in the outpatient clinic control. The application of the scales took 20-25 minutes on average.
- Face-to-face education group (Experimental): Identifying Information Form (IIF), Medication Adherence Report Scale (MARS), and Duke Anticoagulation Satisfaction Scale (DASS) were applied to the face-to-face group in the first interview. They were provided with face-to-face education on the determined date and in the specified environment. At the end of the education, education booklet was given to the individuals. Then, an appointment was made for a month later in hospital environment. In the interview held one month later, the scales were applied again for the last time.
  Interventions: Other: Face-to-face education
- Online education group (Experimental): IIF, MARS, and DASS were also applied to the online education group in the first interview. On the predetermined date and time, online education was given to individuals through video calls held on TEAMS, Google MEET, or WhatsApp. Then, the education booklet was sent to the participants through the application. An appointment date was determined to have another interview a month later. In the interview held a month later, the relevant scales were applied for the last time. At the end of the education, an evaluation was made, and the parts that were seen to be deficient and the issues/questions that the participants raised were repeated. Accordingly, the individuals in both intervention groups were requested to come for control a month later, and the scales were applied for the last time. Education was provided to the participants by the same researcher using the two methods, and the same education content and booklet was used.
  Interventions: Other: Online education

INTERVENTIONS:
Other: Online education — Education content was prepared by the researchers by reviewing the literature. Education content included topics such as oral anticoagulant (OAC) medication introduction, OAC medication use, duration of use, most frequently seen side effects, interaction with other medications and foods, and points to consider while using the medication. While preparing the education content, expert opinions of five nurse academicians were taken. Evaluation of expert opinion was made through the form for Evaluation of the Appropriateness of Printed Materials and Discern. This education content created was provided to the face-to-face and online education groups in one session. Education sessions lasted approximately for 25-30 minutes.
  Arms: Online education group
Other: Face-to-face education — Education content was prepared by the researchers by reviewing the literature. Education content included topics such as OAC medication introduction, OAC medication use, duration of use, most frequently seen side effects, interaction with other medications and foods, and points to consider while using the medication. While preparing the education content, expert opinions of five nurse academicians were taken. Evaluation of expert opinion was made through the form for Evaluation of the Appropriateness of Printed Materials and Discern. This education content created was provided to the face-to-face and online education groups in one session. Education sessions lasted approximately for 25-30 minutes.
  Arms: Face-to-face education group

SUMMARY:
This randomized controlled study was conducted to investigate the effects of face-to-face Education and tele-education given to individuals with atrial fibrillation taking oral Anticoagulants on their medication compliance and satisfaction levels.

The study sample comprised 150 individuals. Of them, 50 were assigned to the control Group, 50 in the experimental group 1, and 50 for the experimental group 2.

Data were collected by the Descriptive Information Form, Medication Compliance Notification Scale and Duke Anticoagulant Satisfaction Scale. The Intervention Group 1 Was given face-to-face education. The Intervention Group 2 was given tele-education.

The control group underwent no intervention.

DETAILED DESCRIPTION:
This randomized controlled study was conducted to investigate effects of face-to-face education and tele-education given to individuals with atrial fibrillation taking oral anticoagulants on their medication compliance and satisfaction levels. The study sample comprised 150 individuals. Of them, 50 were assigned to the control group, 50 to the experimental group 1, and 50 to the experimental group 2. Data were collected with the Descriptive Information Form, Medication Compliance Notification Scale and Duke Anticoagulant Satisfaction Scale. The Intervention Group 1 was given face-to-face education. The Intervention Group 2 was given tele-education.

The control group underwent no intervention. The scales were administered to all the groups twice, at the first and last interviews. Frequency, percentage calculation, Chi-square test, significance test between two means, one-way analysis of variance, Wilcoxon sign test, Fisher test, Bonferroni test and dependent groups t test were used in the analysis of data. The intra-group analysis demonstrated that the Medication Compliance Notification Scale score of the intervention group 1 (face-to-face education group) increased significantly in the final measurement compared to those of the control group and intervention group 2 (tele-education group) (p=.000). The inter-group analysis demonstrated that Duke Anticoagulant Satisfaction Scale scores of the three groups statistically significantly different. The difference stemmed from the intervention group 1.

Face-to-face education given to individuals with atrial fibrillation on oral anticoagulants improved their medication compliance and medication satisfaction levels. Nurses should primarily use face-to-face education in the care and education programs of individuals with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Diagnosed with Atrial fibrillation (AF) for at least a year
* Had been using oral anticoagulant (OACs) for at least 3 months
* Had a smart phone
* Had not previously taken any training on oral anticoagulant medication treatment

Exclusion Criteria:

* The individuals who had disorders that would affect training and experienced complications such as active hemorrhage related to oral anticoagulant use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Identifying Information Form (IIF) | 1 month
  The form developed by the researchers by reviewing the literature consisted of 14 questions regarding the individuals' sociodemographic characteristics (age, gender, marital status, occupation, etc.) and disease characteristics (presence of a chronic disease, etc.)
Medication Adherence Report Scale (MARS) | 1 month
  The 5-point Likert type scale has five items. The total scale score is calculated by summing all item scores. The score to be obtained from the scale ranges between 5-25. High scores obtained from the scale show better medication adherence.
Duke Anticoagulation Satisfaction Scale (DASS) | 1 month
  The 7-point Likert type scale has 25 items under three subscales. High scores obtained from the scale show low medication satisfaction. The highest and lowest scores to be obtained from the scale are 175 and 25, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara bilkent city hospital, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No